CLINICAL TRIAL: NCT00769301
Title: Advancing the Science of Symptom Management and Support for Cancer Patients and Their Caregivers
Brief Title: Symptom Clusters in Cancer Patients and Their Caregivers- a Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Professor, Oslo University Hospital
Other Study IDs: 154-08158d
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2011-06

CONDITIONS: Cancer; Pain; Fatigue; Depression; Sleeping Problems
Keywords: Symptoms; pain; fatigue; depression; sleeplessness; genetic markers; caregiver burden.
MeSH Terms: conditions — Neoplasms; Pain; Fatigue; Depression; Parasomnias; Sleep Initiation and Maintenance Disorders; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA analyses for genotyping subgroups of patients based on their experience with pain, fatigue, sleep disturbance and depression will test the hypothesis that gene polymorphisms within the selected candidate genes will exhibit significant differences in frequency distribution among the different patient subgroups that are identified through cluster analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Not hospitalized cancer patients under active treatment
- 2: Caregivers of these cancer patients

SUMMARY:
The complexity of cancer patients' symptoms and health problems constitutes considerable distress and burden for patients and their family caregivers. To help them manage the illness effectively, there is a need to better understand the complexity of symptoms and symptom clusters in patients and caregivers. Therefore, the purpose of this research is to explore a set of important fundamental research questions to advance the scientific knowledge of cancer patients' and caregivers' symptoms, symptom clusters and health-related quality of life. The investigators will follow 500 cancer patients and their caregivers with repeated measures over 6 months to assess their symptoms, symptom clusters, and quality of life over time. Caregiver burden will also be examined in the caregivers.

DETAILED DESCRIPTION:
The specific aims of the study, where we will follow 500 cancer patients and their caregivers with repeated measures over 6 months, are to:

1. Explore cancer patients' symptoms, symptom clusters and symptom changes over time; and identify subgroups of patients with different symptom clusters.
2. Identify genomic markers for the different patient subgroups.
3. Explore symptoms, symptom clusters and burden in caregivers of cancer patients.
4. Explore relationships between patients' and caregivers' symptoms, symptom clusters, quality of life and caregiver burden.

Patients will be asked to complete questionnaires to collect demographic characteristics and self-reported medical history information, a general symptom inventory, specific measures of the symptoms of pain, sleep disturbance, fatigue, depression, functional status and quality of life. The patients' medical record will be reviewed for disease and treatment information.

The caregivers will also be asked to complete questionnaires about a general symptom inventory, specific measures of the symptoms of pain, sleep disturbance, fatigue, depression, functional status, quality of life and caregiver burden.

Data Analyses will be done to identify symptom clusters of the different symptoms, and to identify patient subgroups based on their symptom experience and quality of life. Variations in symptom clusters and quality of life over time will also be evaluated. Genetic analyses will also be done in the patients.

ELIGIBILITY:
Inclusion Criteria for patients are:

* diagnosed with breast, colon, head and neck or ovarian cancer
* receiving active treatment for their cancer (chemo- or radiation therapy)
* above 18 years of age
* able to read / write /speak Norwegian.

Inclusion criteria for caregivers:

* above 18 years
* read and speak Norwegian
* and written informed consent.

Exclusion Criteria:

* patients who had received radiation on the brain as this may affect their abilities to reliably complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 cancer outpatients (125 with breast cancer and 125 with head and neck cancer receiving radiation therapy and 125 ovarian cancer patients and 125 colon cancer patients receiving chemotherapy)
  and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Physical functioning and quality of life | 5 to 8 times during 6 months

SECONDARY OUTCOMES:
Symptoms will be measured both in patients and caregivers. Caregiver burden will be measured in the caregivers. A blood sample for genetic testing will be taken from the patients once | 5 to 8 times during 6 months for patients. Three times during 6 months for caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Norway (3):
  - Sykehuset Østfold, Fredrikstad
  - Oslo University Hopsital, Rikshospitalet, Oslo
  - Rikshospitalet, Oslo